CLINICAL TRIAL: NCT02278770
Title: Pilot Study: MRI Study of Diverticular Disease Symptoms and Its Relationship to Visceral Adipose Tissue
Brief Title: DD Obesity MRI Study
Acronym: DDOMRI
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 10/H0405/80
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Diverticular Disease
Keywords: diverticular disease; MRI; visceral and subcutaneous fat; adipokines
MeSH Terms: conditions — Diverticular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and stool
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, our novel MRI techniques for studying the small bowel will be applied to patients with diverticular disease. The ratio of visceral to subcutaneous fat will also be determined using MRI measurements. These data will be correlated with measurements of adipokines to determine if visceral fat has a specific influence on the severity of diverticular disease.

DETAILED DESCRIPTION:
Colonic diverticulosis is the most common structural abnormality of the colon and studies suggest that its incidence and/or complications are increasing. Increasing evidence suggests a link between obesity and complications of diverticular disease. With the prevalence of obesity increasing in westernised populations, the risk of complications from diverticular disease is likely to also increase. At present however, there is little understanding of how diverticular complications are increased by obesity. A high BMI might be a surrogate marker for other lifestyle factors which predispose to diverticular complications. Visceral fat may also have an influence on related complications, due to the compounds secreted by adipocytes.

Altered bowel habit is a common complaint of diverticular patients. The cause is not well understood, is probably multi-factorial, and may include changes in the small bowel. Until recently, studies of the large and small bowel required intestinal intubation and perfusion and could not be performed on the undisturbed colon. New MRI techniques have now been developed, which allow these areas to be studied non-invasively. Abdominal fat can also be measured using MRI, and the distribution of subcutaneous and visceral fat will be compared for symptomatic and asymptomatic diverticular patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have symptomatic and asymptomatic Diverticular disease confirmed on colonoscopy, barium enema or CT scan (Symptomatic disease is defined as lower abdominal pain >1hr on 3 or more days per month for longer than 3 months.)

Exclusion Criteria:

* 1. Pregnant or lactating women. 2. Severe co-morbidity; e.g. heart failure, respiratory failure, alcoholism or drug dependence, 3. Inability to give informed consent. 4. If the participant has taken part in any other study on campus in the last 3 months they will not be able to take part in this study.

  5. Inability to lie supine 6. Inability to stop laxatives for 24hrs and antispasmodics or ondansetron for 8 hours prior to the commencement of the MRI study.

  7. Using long-term NSAIDs (non-steroidal anti-inflammatory agents e.g. ibuprofen), antibiotics or immunosuppressant drugs 8. Antibiotics within last 3 months 9. Other gastrointestinal inflammatory problems e.g. ulcerative colitis, Crohn's or Coeliac disease

MRI exclusions 10. Have a metallic implant 11. Have shrapnel inside the body 12. Ever had metallic fragments in the eye 13. Claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include:
  1. Participants with symptomatic DD stratified by patient heath questionnaire 12 somatic symptom scale
  2. Participants with asymptomatic DD
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Difference in the volume of visceral fat compared to abdominal subcutaneous fat between symptomatic and asymptomatic DD groups | 3 years

SECONDARY OUTCOMES:
Adiponectin and leptin serum levels between symptomatic and asymptomatic DD groups | 3 years
The incidence of diarrhoea between participants with a BMI <25kg/m2 and those >25kg/m2 | 3 years
Adiponectin and leptin serum levels between DD groups with and without diarrhoea | 3 years
Small and large bowel water and lumen diameter in symptomatic and asymptomatic DD groups | 3 years
Calprotectin levels between symptomatic and asymptomatic DD groups | 3 years
Microbiological gut profile between symptomatic asymptomatic DD groups | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robin C Spiller, MD, FRCP, Study Chair — Nottingham University Hospitals; Jan K Smith, Principal Investigator — Nottingham University Hospitals; David J Humes, Principal Investigator — Nottingham Unversity Hospitals; Luca Marciani, Principal Investigator — Nottingham University Hospitals